CLINICAL TRIAL: NCT06764394
Title: The Effect of Myofascial Release Exercises on Viscoelastic Changes of the Pectoralis Major Muscle
Brief Title: The Effect of Myofascial Release Exercises on Viscoelastic Changes of the Pectoralis Major Muscle, Pain, Range of Motion and Shoulder Functionality in Individuals Receiving Adjuvant Radiotherapy After Breast Cancer Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Acibadem University (Other)
Responsible Party: Principal Investigator, Özlem Feyzioğlu, Asistant professor, Acibadem University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ATADEK 2024-19/733
Record Dates: First submitted 2025-01-02; First posted 2025-01-08 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-01

CONDITIONS: Breast Cancer
Keywords: myofascial release exercises, breast cancer, radiotherapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- home based exercise group (Active Comparator): home-based exercise 5 days a week
- Myofascial release exercise group (Experimental): home based exercise plus Myofascial release exercise
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — home based exercise 5 days/week
  Other Names: home based exercise
Other: Exercise — home based exercise plus myofacial release exercise Myofascial release exercises will continue for 6 weeks, 2 sessions per week and each session will continue for 30 minutes.All evaluations will be performed at the beginning of radiotherapy treatment and at the end of the 6th week.
  Arms: Myofascial release exercise group

SUMMARY:
Chemotherapy, hormone therapy and radiotherapy used in the treatment of breast cancer try to prevent the recurrence of cancer. In addition to the benefits of radiotherapy, such as a decrease in recurrence and an increase in long-term survival, it may have side effects that may affect the well-being and daily life activities of patients. One of the treatment modalities used to cope with treatment-related side effects is myofascial release exercises. Myofascial release exercises can help reduce adhesions caused by scar tissue and fibrosis caused by radiation. In the literature, there is no study investigating the effect of myofascial release exercises on pectoralis major muscle viscoelastic structure. For this purpose, our study aims to investigate the effect of myofascial release exercises performed in addition to home exercise programme on pectoralis major muscle viscoelastic structure, pain, range of motion and shoulder functionality.

ELIGIBILITY:
Inclusion Criteria:

* -Stage I-II-III defined by radiation oncologists after breast cancer surgery and who will start radiotherapy
* Breast conserving surgery or total mastectomy with axillary lymph node dissection during surgery
* No neurological or orthopaedic problems that may limit the range of motion of the shoulder joint in the preoperative evaluations,
* Individuals who volunteer to participate in the study will be included.

Exclusion Criteria:

* Previous breast clamp surgery on the same side or contralateral side,
* With a metastatic cancer focus,
* Post-surgical resistance, infection and open wound, pacemaker,
* Patients with a Mini Mental State Examination test score of less than 21 will be excluded from the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-12-20 (Actual); Primary Completion 2025-03-30 (Actual); Study Completion 2025-05-10 (Actual)

PRIMARY OUTCOMES:
Tone - pectoralis major | 6 weeks
  Myoton® PRO (Myoton Ltd, Myoton AS, Estonia) device will be used to objectively evaluate the measurement of Pectoralis Major muscle tone of the patients who will participate in the study. Myoton® PRO is a portable digital device that measures the tone with an objective and noninvasive method.
  A constant pre-pressure (0.18 N) is applied to the skin surface to compress the subcutaneous superficial tissues. The tension state of the tissue that characterized by the natural oscillation frequency; Hz.
Range of motion | 6 weeks
  Shoulder range of motion will be evaluated by digital goniometer. Shoulder flexion degree, shoulder extension degree, abduction and adduction degree, internal rotation and external rotation degree will be assessed with digital goniometer. The results will be recorded in degrees.

SECONDARY OUTCOMES:
Pain - Visual Analogue Scale | 6 weeks
  Visual Analogue Scale is one of the simple and common methods used in pain assessment. Self reported pain intensity during the rest and the activity measured by 0-10 centimeter chart. Visual Analogue Scale (VAS), where 0 indicates no pain or best and 10 indicates the most intense pain imaginable or worst. The patient will mark the severity of the pain on a 10 cm long chart
Shoulder Pain and Disability Index- SPADI | 6 weeks
  Shoulder Pain and Disability Index: The Shoulder Pain and Disability Index (SPADI) is used to assess the pain and disability of individuals during certain activities. The SPADI is an assessment method consisting of two sub-headings, pain and functional status, which are completed in approximately 5-10 minutes. The first part consists of 5 questions to assess the level of pain during lying down, lying on the affected side and pushing activities. The second part consisting of 8 questions evaluates the functional status by questioning dressing, personal care and carrying activities. The subjects answer each question using a 10 cm Visual Analogue Scale. The answers to the questions are calculated as percentiles. The total score varies between 0-130, with the higher percentile indicating increased disability.
Quality of Life- Functional Assessment of Cancer Therapy-Breast" (FACT-B) | 6 weeks
  It is designed to evaluate the quality of life in breast cancer patients from multiple perspectives. Its validity and reliability have been demonstrated. It consists of 5 subscales that assess quality of life as physical condition (7 questions), social life and family status (7 questions), emotional status (6 questions), activity status (7 questions), and other breast cancer-specific concerns (9 questions). The survey has 5-point likert scoring (0=not at all, 1=a little, 2=a little, 3=quite a lot, 4=a lot) . The total score is calculated by summing the subscale scores. A higher score on the questionnaire indicates a higher quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- SBU. Prof. Dr. Cemil Taşçıoğlu City Hospital- Oncology Clinic, Istanbul, Turkey (Türkiye)